CLINICAL TRIAL: NCT04342676
Title: Lymph Node Ratio and Kras Mutation in Risk Stratification of Colon Cancer
Brief Title: Lymph Node Ratio and Kras Mutation in R Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 20202
Record Dates: First submitted 2020-04-03; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Colon Cancer Stage III
MeSH Terms: conditions — Colonic Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- patients (Experimental): LNR measured by (number of metastatic lymph nodes/total number of lymph nodes excised). and K ras (polymerase chain reaction (PCR) and pyrosequencing targeted for KRAS codons 12-13 was performed )
  Interventions: Device: k ras; Drug: Panitumumab

INTERVENTIONS:
Device: k ras — K ras
Drug: Panitumumab — vectibex in stage iv
  Other Names: vectibex

SUMMARY:
clinical impact of LN ratio with Kras expression in colon cancer

DETAILED DESCRIPTION:
LNR and K ras were evaluated with correlated with different clinicopathological parameters of the patients, PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

* Stage III colon cancer

Exclusion Criteria:

* Stage I, II, IV

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
LNR and K ras were evaluated with correlated with different clinicopathological parameters (Gender, CEA, tumor size, tumor grade and response to treatment). | 2 years
  impact on response

SECONDARY OUTCOMES:
LNR and K ras were evaluated and ASSOCIATION with PFS and OS. | 2 years
  impact on survival

CONTACTS AND LOCATIONS:
Overall Officials: Tawfik A Elkhodary, MD, Study Chair — Oncology Center Mansoura University
Locations (1):
- Mansoura University Oncology Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
after publication